CLINICAL TRIAL: NCT05329233
Title: Continuous ORI Monitoring is a Non-invasive Monitoring Method
Brief Title: Comparison of the Effects of High, Low and Minimal Flow Anesthesia Managements on ORI and Partial Oxygen Pressure
Status: Completed | Type: Observational
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Hale Kefeli Celik, Anesthesiologist, Samsun Education and Research Hospital
Other Study IDs: KAEK-2020/1/1
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: General Anesthetic
Keywords: low flow anesthesia; oxygen reserve index; arterial oxygen pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- minimal flow: For minimal-flow anesthesia, oxygen 0.3 L/min and medical air 0.2 L/min (FGF 0.5 L/min, FiO2 68%) were administered to patients in group M.
  Interventions: Device: Masimo Radical-7 Pulse CO-Oximeter
- low flow: For low-flow anesthesia, oxygen 0.37 L/min and medical air 0.63 L/min (FGF 1 L/min, FiO2 50%) were administered to patients in group L.
  Interventions: Device: Masimo Radical-7 Pulse CO-Oximeter
- high flow: For high-flow anesthesia, oxygen 1 L/min and medical air 3 L/min (FGF 4 L/min, FiO2 40%) were administered to patients in group H.
  Interventions: Device: Masimo Radical-7 Pulse CO-Oximeter

INTERVENTIONS:
Device: Masimo Radical-7 Pulse CO-Oximeter — The Masimo Radical-7 Pulse CO-Oximeter is a device for the measurement of pulse oximetry, oxygen reserve index (ORi), perfusion index (PI), and pleth variability index (PVI). The device is the product of a company called Masimo Inc, Irvine, CA, USA

SUMMARY:
The aim of our study is to show that continuous oxygen reserve index monitoring is a non-invasive monitoring method that can be used as a supporting parameter to PaO2 in blood gas in hypoxia and hyperoxia monitoring when different fresh gas flow is used in general anesthesia.

DETAILED DESCRIPTION:
Ninety patients included in the study were classified into three groups. After the high flow period, FGF and inspired oxygen fraction (FiO2) was set to be 4 L/m and 40% in group H (high flow), 1 L/m and 50% in group L (low flow) and 0.5 L/m and 68% in group M (minimal flow), respectively.

Patients were transferred into the operating room, monitored and premedication with 0.03 mg/kg of midazolam was administered. Subsequently, the right radial artery was cannulated under local anesthesia and basal blood samples were taken. After preoxygenation (100% O2, 6 L/min, 3 min.), anesthesia induction was performed with intravenous administration of 40-60 mg lidocaine, 2 mg/kg propofol, 0.6 mg/kg rocuronium and 1.5 mcg/kg fentanyl. Patients were ventilated in volume-controlled mode (Dräger Perseus® A500 Anaesthesia Workstation, Dräger, Germany) that allows continuous monitorization of airway pressure, exhaled gas volume, FiO2, volatile anesthetic substance concentration, and CO2 concentration within the scope of the Common European Standard EN 740. Medical air was used as the carrier gas. End-tidal carbon dioxide (EtCO2) was continuously monitored after intubation, and tidal volume and ventilation rates were adjusted to maintain EtCO2 at 30-40 mmHg. In maintenance, general anesthesia was provided in all three groups by inhalation of remifentanil 0.05-0.2 mcg/kg/min and FGF 4 L/min 50% oxygen-medical air mixture with 6-8% desflurane. After intubation, 6% desflurane was administered with a fresh gas flow of 4 L/min for 10 minutes in all three groups, and the MAC value was adjusted to 1.

Thereafter, oxygen 1 L/min, and medical air 3 L/min (FGF 4 L/min, FiO2 40%) were administered to patients in group H for high-flow anesthesia; oxygen 0.37 L/min, medical air 0.63 L/min (FGF 1 L/min, FiO2 50%) to patients in group L for low-flow anesthesia; oxygen 0.3 L/min and medical air 0.2 L/min (FGF 0.5 L/min, FiO2 68%) to patients in group M under minimal flow anesthesia. After reaching adequate MAC values after 10 minutes of intubation, FiO2 was reduced to 40% in Group H, keeping the FGF unchanged; in Group L fresh gas flow was reduced to 1 L/min, in Group M fresh gas flow was reduced to 0.5 L/min, and the scale setting of desflurane was adjusted in order to achieve MAC 1 for the remainder of the surgery.

A disposable sensor (RD Rainbow Lite Set ORI Probe, Masimo Corp. Irvine CA), shielded from light, was placed on the left index finger to record the data displayed with Masimo Radical 7 pulse CO-Oximeter (Masimo Corp. Irvine CA).

At the end of the surgical procedure in all patients, the vaporizer was turned off and high FGF (4 L/min, FiO2 100%) was applied to ensure rapid removal of the anesthetic gases from the lungs, and manual ventilation was started. Sugammadex (2-4 mg/kg iv.) was administered to reverse the residual muscle relaxation at the end of the operation in patients who did not experience complications during the operation, and after spontaneous breathing was achieved, the patients were extubated in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* ASA II and III patients,
* Aged between 18-75 years,
* who were scheduled to undergo elective open abdominal surgery lasting <60 minutes under general anesthesia

Exclusion Criteria:

* refusal of consent to study inclusion by the patient or his/her guardian,
* inability to use the sensor due to finger deformation or hypoperfusion,
* having a history of malignant hyperthermia,
* presence of clinically significant anemia, morbid obesity, alcohol or drug addiction, having a severe cardiac, renal or hepatic impairment,
* having a history of cerebrovascular disease,
* being a pregnant or presently lactating and having local anesthetic or opioid sensitivity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA II and III patients aged between 18-75 years, who were scheduled to undergo elective open abdominal surgery lasting <60 minutes under general anesthesia
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
The use of continuous ORI monitoring as a supporting parameter to PaO2 in blood gasses during hypoxia and hyperoxia | intraoperative period
  To show that continuous ORI monitoring is non-invasive monitoring that can be used as a supporting parameter for PaO2 in blood gas in hypoxia and hyperoxia monitoring when different fresh gas flows (4, 1, 0.5 L/min) are used in general anesthesia practice.

SECONDARY OUTCOMES:
The use of continuous ORI monitoring as a supporting parameter to PaO2 in blood gasses during hypoxia and hyperoxia | İntraoperative period
  Parameters were recorded at nine time frames: T1 (5 minutes before anesthesia induction), T2 (after intubation), T3 (at the start of 0.5-1-4 L/min), T4 (at the 10th minute of low flow), T5 (at the 30th minute of low flow), T6 (at the 60th minute of low flow), T7 (at the 90th minute of low flow), T8 (at the 120th minute of low flow), T9 (at the end of the surgery, ventilation with 100% oxygen) and T10 (5 min after extubation).

CONTACTS AND LOCATIONS:
Overall Officials: Zahide Doganay, Professor, Study Chair — Samsun Research and Education Hospital
Locations (1):
- Samsun Research and Education Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Our data and statistical analysis of each investigated all parameter and data are available after the publication of the clinical study
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after the publication of our data upon request from the researchers.
Access Criteria: There is no internet website to obtain data but the researchers can contact Dr. Naci Murat, Ondokuz Mayis University, Samsun, Turkey.

REFERENCES:
- [Result] Baxter AD. Low and minimal flow inhalational anaesthesia. Can J Anaesth. 1997 Jun;44(6):643-52; quiz 652-3. doi: 10.1007/BF03015449. PMID 9187785
- [Result] Vos JJ, Willems CH, van Amsterdam K, van den Berg JP, Spanjersberg R, Struys MMRF, Scheeren TWL. Oxygen Reserve Index: Validation of a New Variable. Anesth Analg. 2019 Aug;129(2):409-415. doi: 10.1213/ANE.0000000000003706. PMID 30138170
- [Result] Scheeren TWL, Belda FJ, Perel A. The oxygen reserve index (ORI): a new tool to monitor oxygen therapy. J Clin Monit Comput. 2018 Jun;32(3):379-389. doi: 10.1007/s10877-017-0049-4. Epub 2017 Aug 8. PMID 28791567